CLINICAL TRIAL: NCT06590129
Title: Effectiveness in Functional Recovery and Pain Reduction Following Hydrodissection vs Rehabilitation in Patients With Carpal Tunnel Syndrome
Brief Title: Functional Recovery and Pain Reduction Post-hydrodissection vs Rehabilitation in Patients With Carpal Tunnel Syndrome (Hydrocarpal)
Acronym: hydrocarpal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Roberto Carlos Pech Arguelles, Director of Research, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-2023-3201-068
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Carpal Tunnel Syndrome (CTS)
Keywords: Carpal Tunnel Syndrome; Rehabilitation; physical therapy; Hidrodissection; Physiotherapy; Median nerve neuropathy
MeSH Terms: conditions — Carpal Tunnel Syndrome; Median Neuropathy | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Prospective, longitudinal, randomized clinical study, including 50 patients diagnosed with CTS. Two groups were compared: one received physical therapy and the other received median nerve ultrasound guided hydrodissection plus physiotherapy evaluated initially, 4 and 12 weeks with the Boston questionnaire and the Visual Analogue Scale (VAS).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Only Rehabilitation (Active Comparator): Evaluated with the Boston questionnaire and the Visual Analogue Scale (VAS), then te patients were enroled to a 15-20 sessions in rehabilitation area with physical media: paraffin glove (10 coats for 15min), mobilizations of wrist and fingers, strectching of wrist and fingers tendons/muscles, muscle stregthening whit isometric or isotonic excercises to intrinsic muscles of the hand an forearm, and occupational therapy with techniques for sensory return, nerve and tendon sliding techniques, activities aimed at improving basic hand functions and work simulation activities.
  Interventions: Other: Physiotherapy
- Median nerve ultrasound guided hidrodissection + rehabilitation (Experimental): Evaluated with the Boston questionnaire and the Visual Analogue Scale (VAS), then an ultrasound guided hidrodissection of the median nerve with 4.5ml of glucosade solution was performed.
  The patients were enrolled into 15-20 sessions in rehabilitation área with the same protocolo of the control group.
  Interventions: Procedure: hydrodissection of median nerve; Other: Physiotherapy

INTERVENTIONS:
Procedure: hydrodissection of median nerve — Ultrasound guided hydrodissection of median nerve in carpal tunnel with 5% dextrose solution
  Arms: Median nerve ultrasound guided hidrodissection + rehabilitation
Other: Physiotherapy — 5-20 sessions in rehabilitation area with physical media: paraffin glove (10 coats for 15min), mobilizations of wrist and fingers, strectching of wrist and fingers tendons/muscles, muscle stregthening whit isometric or isotonic excercises to intrinsic muscles of the hand an forearm, and occupational therapy with techniques for sensory return, nerve and tendon sliding techniques, activities aimed at improving basic hand functions and work simulation activities.

SUMMARY:
This study pretend to evaluate the effectiveness of hydrodissection vs only rehabilitation in improving pain and function in patients with CTS.

DETAILED DESCRIPTION:
This prospective, longitudinal, randomized in two groups clinical study pretend to evaluate the effectiveness of hydrodissection vs only rehabilitation in improving pain and function in patients with CTS, evaluated initially and at 4 and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* men and women ≥18 years of age,
* members referred to and treated at the Physical Medicine and Rehabilitation Service of HGR N°1, IMSS Mérida Yucatán, and who had a clinical or electrophysiological diagnosis of carpal tunnel syndrome.

Exclusion Criteria:

* included a clinical or electrophysiological diagnosis of radiculopathy, plexopathy, polyneuropathy, or other peripheral neuropathy;
* current diagnosis of cancer, coagulopathy, thoracic outlet syndrome;
* active infectious process or current fracture in the thoracic limb;
* previous surgery for carpal tunnel release;
* inability to cooperate with filling out scales, physical examination, or infiltration, as clearly detailed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Function | Initially, 4 and 12 weeks.
  Boston´s carpal tunnel questionnaire results, where each item is scored from 1 (no symptoms/difficulties) to 5 (the worst symptoms/cannot perform the activity at all). The mean score for each scale is calculated, resulting in a score between 1 and 5, with higher scores indicating worse symptoms or function.
Pain | Initially, 4 and 12 weeks.
  Visual Analogue Scale (VAS) is a pain intensity measurement tool that uses a 10 cm line with two end points to indicate no pain and worst possible pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Regional No.1 "Lic. Ignacio García Téllez" IMSS, Calle 41 101, Fénix, 97155 Mérida, Yuc., Mérida, Yucatán, Mexico

IPD SHARING:
Plan to Share IPD: No
All IPD collected throughout the trial, only IPD used in the results publication

REFERENCES:
- [Background] Lin CP, Chang KV, Huang YK, Wu WT, Ozcakar L. Regenerative Injections Including 5% Dextrose and Platelet-Rich Plasma for the Treatment of Carpal Tunnel Syndrome: A Systematic Review and Network Meta-Analysis. Pharmaceuticals (Basel). 2020 Mar 18;13(3):49. doi: 10.3390/ph13030049. PMID 32197544
- [Background] Shen YP, Li TY, Chou YC, Ho TY, Ke MJ, Chen LC, Wu YT. Comparison of perineural platelet-rich plasma and dextrose injections for moderate carpal tunnel syndrome: A prospective randomized, single-blind, head-to-head comparative trial. J Tissue Eng Regen Med. 2019 Nov;13(11):2009-2017. doi: 10.1002/term.2950. Epub 2019 Aug 20. PMID 31368191
- [Background] Wu YT, Ho TY, Chou YC, Ke MJ, Li TY, Tsai CK, Chen LC. Six-month Efficacy of Perineural Dextrose for Carpal Tunnel Syndrome: A Prospective, Randomized, Double-Blind, Controlled Trial. Mayo Clin Proc. 2017 Aug;92(8):1179-1189. doi: 10.1016/j.mayocp.2017.05.025. PMID 28778254
- [Background] Neo EJR, Shan NT, Tay SS. Hydrodissection for Carpal Tunnel Syndrome: A Systematic Review. Am J Phys Med Rehabil. 2022 Jun 1;101(6):530-539. doi: 10.1097/PHM.0000000000001846. Epub 2021 Jul 14. PMID 34261895
- [Background] Wu YT, Chen YP, Lam KHS, Reeves KD, Lin JA, Kuo CY. Mechanism of Glucose Water as a Neural Injection: A Perspective on Neuroinflammation. Life (Basel). 2022 Jun 2;12(6):832. doi: 10.3390/life12060832. PMID 35743863
- [Background] Kjeken I, Sundin U. Management of carpal tunnel syndrome in primary care. Rheumatology (Oxford). 2023 Feb 1;62(2):495-496. doi: 10.1093/rheumatology/keac396. No abstract available. PMID 35894646
- [Background] Burton CL, Chesterton LS, Chen Y, van der Windt DA. Clinical Course and Prognostic Factors in Conservatively Managed Carpal Tunnel Syndrome: A Systematic Review. Arch Phys Med Rehabil. 2016 May;97(5):836-852.e1. doi: 10.1016/j.apmr.2015.09.013. Epub 2015 Oct 9. PMID 26440776
- [Background] Genova A, Dix O, Saefan A, Thakur M, Hassan A. Carpal Tunnel Syndrome: A Review of Literature. Cureus. 2020 Mar 19;12(3):e7333. doi: 10.7759/cureus.7333. PMID 32313774
- [Background] Thiese MS, Gerr F, Hegmann KT, Harris-Adamson C, Dale AM, Evanoff B, Eisen EA, Kapellusch J, Garg A, Burt S, Bao S, Silverstein B, Merlino L, Rempel D. Effects of varying case definition on carpal tunnel syndrome prevalence estimates in a pooled cohort. Arch Phys Med Rehabil. 2014 Dec;95(12):2320-6. doi: 10.1016/j.apmr.2014.08.004. Epub 2014 Aug 28. PMID 25175160
- [Background] Lores Peniche JA, Huchim Lara O, Méndez-Domínguez N. Carpal Tunnel Syndrome: Epidemiological Analysis of Cases Treated in Hospital Services in Mexico. Physiotherapy. 2020;42(2):69-74.
- See also: Carpal tunnel syndrome: Treatment and prognosis [Internet]. UpToDate — https://www.uptodate.com/contents/carpal-tunnel-syndrome-treatment-and-prognosis
- See also: Surgery for carpal tunnel syndrome [Internet]. UpToDate. — https://www.uptodate.com/contents/surgery-for-carpal-tunnel-syndrome